CLINICAL TRIAL: NCT01520584
Title: Vitamins ,Minerals and Amino Acids Supplement Intake in Infertile Men;the Effect on Sperm Parameters,Fertilization Rate and Embryo Quality. A Double Blind Randomized Controlled Trial
Brief Title: Supplement Intake in Infertile Men;the Effect on Sperm Parameters,Fertilization Rate and Embryo Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 0103-10
Record Dates: First submitted 2012-01-14; First posted 2012-01-30 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Oligospermia
MeSH Terms: conditions — Oligospermia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamale (Active Comparator)
  Interventions: Dietary Supplement: Vitamale
- sham pill (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamale

INTERVENTIONS:
Dietary Supplement: Vitamale — men will receive the vitamale dietary supplement compared to a sham pill
  Other Names: amino acid minerals and vitamin supplement

SUMMARY:
The vitamin,minerals and amino acid supplementation for 3 months will improve the semen parameters,fertilization rate and embryo quality in subfertile men undergoing IVF treatment

DETAILED DESCRIPTION:
With the supplement intake containing amino acids, vitamins and minerals designed to improve sperm parameters, the couples undergoing IVF treatment will benefit as the change and improvement of sperm parameters will increase the fertilization rate and improve the embryo quality thus allowing shorter time for pregnancy achievement and less frustration with long duration of treatments

ELIGIBILITY:
Inclusion Criteria:

* healthy male age 20-50
* at least one IVF cycle without pregnancy
* sperm parameters:
* Oligospermia 5-20*106
* Teratospermia 6-14% normal forms
* Asthenospermia <30% motility

Exclusion Criteria:

* female factor infertility
* age > 50 or under 20
* testicular problem on physical examination
* history of malignancy and /or chemotherapy
* usage of antiandrogen/testosterone
* history of drug abuse/alcohol
* a known endocrinological problem
* current STD or genitourinary infection
* Retrograde Ejaculation
* Y chromosome microdeletion
* Karyotype abnormalities

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Sperm parameters | 3 months of treatment
  Men suffering from a "male factor" problem and after one failed IVF treatment will be given the supplement for 3 months after which the sperm parametrs will be evaluated and compared to pre-supplement data and later the embryo quality and fertilization rate will reviewed analyzed and compared

CONTACTS AND LOCATIONS:
Overall Officials: Dana Irge, DR, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

REFERENCES:
- [Derived] de Ligny W, Smits RM, Mackenzie-Proctor R, Jordan V, Fleischer K, de Bruin JP, Showell MG. Antioxidants for male subfertility. Cochrane Database Syst Rev. 2022 May 4;5(5):CD007411. doi: 10.1002/14651858.CD007411.pub5. PMID 35506389